CLINICAL TRIAL: NCT00374881
Title: A Randomized, Double-Blind, Single-Center, 5 Way Cross-Over Study to Assess the Effect of Adding Oral Phenylephrine and Oral Sorbitol to Low Dose (1.5 mg) Plain Oral Morphine in Human Volunteers: Analgesia and Side Effect Assessment.
Brief Title: A Study of the Safety and Efficacy of Combination Therapy With Morphine, Phenylephrine and Sorbitol in Human Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioLineRx, Ltd. (Industry)
Responsible Party: BioLineRx, BioLineRx
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: BL-3010
Record Dates: First submitted 2006-09-11; First posted 2006-09-12 (Estimated); Last update posted 2008-04-15 (Estimated); Status verified 2008-04

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Active Comparator): Morphine High Dose
  Interventions: Drug: Morphine
- 2 (Placebo Comparator): Morphine Low Dose
  Interventions: Drug: Morphine
- 3 (Placebo Comparator): Sorbitol Phenylephrine
  Interventions: Drug: Sorbitol+Phenylephrine
- 4 (Experimental): Sorbitol high concentration+Phenylephrine+Morphine
  Interventions: Drug: Sorbitol+Phenylephrine+Morphine
- 5 (Experimental): Sorbitol low concentration+Phenylephrine+Morphine
  Interventions: Drug: Sorbitol low concentration+Phenylephrine+Morphine

INTERVENTIONS:
Drug: Morphine — Morphine
  Arms: 1
Drug: Morphine — Morphine low dose
  Arms: 2
Drug: Sorbitol+Phenylephrine — Sorbitol+Phenylephrine
  Arms: 3
Drug: Sorbitol+Phenylephrine+Morphine — Sorbitol+Phenylephrine+Morphine
  Arms: 4
Drug: Sorbitol low concentration+Phenylephrine+Morphine — Sorbitol low concentration+Phenylephrine+Morphine
  Arms: 5

SUMMARY:
Efficacy and Safety of the combined oral adjuvants phenylephrine and sorbitol on oral low dose morphine analgesia.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the efficacy of the combined oral adjuvants phenylephrine and sorbitol on oral low dose morphine analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent
* Healthy male or female between 18 and 40 years of age, inclusive.
* Women have to test negative for pregnancy.
* Body weight within 15% of ideal body weight based on Metropolitan Life assurance tables.
* No concomitant medications (prescription, OTC, vitamins, dietary supplements) within 7 days prior to administration of study medication and during the study period.
* Ability to adhere to the visit schedule and protocol requirements and be available to complete the study
* Ability to participate successfully in training sessions that will be arranged for the volunteers prior to the study day, during which they will acquire consistency in the tests to be performed.
* Ability to satisfy a medical examiner about fitness to participate in the study

Exclusion Criteria:

* prior use of chronic opioids
* mental illness prior or present
* evidence of significant concomitant disease, including renal, hepatic, cardiovascular, pulmonary, endocrinological, hematopoietic, or gastrointestinal disease, a neoplasm or any other clinically significant medical disorder, which in the Investigator's judgment contraindicate administration of the study medications
* known allergy to any of the drugs used in this study
* history of drug or alcohol abuse
* significant abnormalities in screening physical exam
* administration of drugs that may potentially inhibit or induce liver cytochrome P450 activity within 3 weeks prior to Day 0
* any acute medical situation (e.g. acute infection) within 48 hours of Day 0, which is considered of significance by the Principal Investigator
* unusual diet
* administration of experimental medications within the previous 12 weeks.
* inability to communicate well with the Investigator (i.e., language problem, poor mental development or impaired cerebral function)
* subjects who, in the judgment of the investigators, are likely to be non-compliant or uncooperative or unwilling to sign a consent form

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2006-09; Primary Completion 2007-06 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Safety | 8 hours

SECONDARY OUTCOMES:
Efficacy | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Yehuda Ginosar, Bsc, MBBS, Principal Investigator — Department of Anesthesiology, Hadassah Hebrew University Medical Center
Locations (2):
- Israel (2):
  - Hadassah Hebrew University Medical Center, Department of Anesthesiology, Jerusalem
  - Hadassah En Kerem Medical Centre, Jerusalem